CLINICAL TRIAL: NCT00877721
Title: Self Mobility Improvement in the Elderly by Counteracting Falls (SMILING)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: European Union (Other)
Responsible Party: Itshak Melzer PhD, PT, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SOR483209CTIL; MZ4832
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2009-04

CONDITIONS: Falls
Keywords: Postural Control; Gait; Falls; Elderly; Old adults (65 years old and older) with low risk of falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- balance treatment (Experimental)
  Interventions: Device: Self Mobility Improvement in the eLderly by using the SMILING system

INTERVENTIONS:
Device: Self Mobility Improvement in the eLderly by using the SMILING system — The effect of treatment with the SMILING system on postural stability and gait of elderly individuals will be measured using RCT cross over study design

SUMMARY:
Experimental design overview:

The proposed project is a prospective experimental study design. Independent old adults (age 65 years old and older) who suffer from minor balance problems willing to participate in the study will be tested with well-established measuring techniques of balance and gait before and 4 weeks after balance training program using the "Self Mobility Improvement in the Elderly by Counteracting Falls" system (SMILING system). The study design is randomized clinical trial (RCT), cross over, single blinded study design where 30 subjects will randomly be allocated into experimental or control groups that will switch groups after 4 weeks of intervention.

Random sequence generation will be performed by a staff member who will not interact with subjects during the balance-testing sessions. Subjects will be informed that they are to be randomly assigned to one of the two groups, both receiving gait training program.

The staff member who administers the training programs will be the only member of the research team aware of the subjects' group allocations.

A 'blinded' research assistant will administer the balance tests and will perform any data processing that involves subjective judgments.

Scripts will be used during testing to ensure that all subjects receive the same instructions.

Testing session between two training periods (T1) will take one week.

ELIGIBILITY:
The inclusion criteria are:

Self-reported information

1. age ≥ 65 years,
2. able to walk at least 20 meters independently, i.e., without personal assistance and without an assistive device, except for a single point cane
3. one or more falls in the previous year (falls during sport activities excluded).

Standardized physical and cognitive functional tests

1. Tinetti's POMA score below 26 (strictly)
2. MMSE test with score ≥ 24
3. GDS test with score <10

The exclusion criteria are:

1. Self-reported information
2. age < 65 years
3. inability to walk 20 meters safely (self-report) or walk with personal assistance or with an assistive device (except single point cane for fallers)
4. inability to recall fall status in the previous year
5. severe visual impairment (e.g., impaired ability to read, watch TV, or drive a car)
6. severe hearing impairment (e.g., unable to follow a conversation, to use a phone)
7. Standardized physical and cognitive functional tests
8. Tinetti's POMA score less than 19
9. MMSE score < 24
10. GDS test with score ≥ 10
11. Medical conditions (filled in by the family doctor of the subject)
12. wearing a pacemaker, a cardiac defibrillator or any other electronic implant
13. severe gait impairment precluding safe walking over 20 meters due to:
14. focal lower limb muscle weakness or palsy (e.g., unable to raise leg/foot from floor)
15. neurological diseases, including diseases such as severe Parkinson's disease, Multiple Sclerosis, status post stroke with hemi-syndroma, cervical or lumbar stenosis with compression myelopathy, polyneuropathy with severe proprioceptive impairment, Menier
16. severe cardiovascular disease
17. foot problems, lower limb amputation or joint arthrodesis
18. terminal diseases (defined as estimated life expectancy of less than 6 months).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
gait analysis | time 1: pre test; time 2 post test (4 weeks after pre test) and time 3 follow up (8 weeks after pre test)

SECONDARY OUTCOMES:
Tinetti's performance-oriented mobility assessment (POMA score), CODEX test, GDS test | time 1: pre test; time 2 post test (4 weeks after pre test) and time 3 follow up (8 weeks after pre test)
CODEX test | time 1: pre test; time 2 post test (4 weeks after pre test) and time 3 follow up (8 weeks after pre test)
GDS test | time 1: pre test; time 2 post test (4 weeks after pre test) and time 3 follow up (8 weeks after pre test)

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Grinshpon, MD, Study Chair — Soroka University Medical Center; Itshak Melzer, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- SorokaUMC, Beersheba, Israel